CLINICAL TRIAL: NCT05292417
Title: A Trial of Hypofractionation Radiotherapy in Combination With Sintilimab，GM-CSF and Fruquintinib in Patients With MSS Metastatic Colorectal Carcinoma (mCRC)
Brief Title: Radiotherapy in Combination With Sintilimab，GM-CSF and Fruquintinib in Patients With MSS mCRC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Caimingquan
Record Dates: First submitted 2022-03-10; First posted 2022-03-23 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Radiation Dose Hypofractionation; Radiotherapy; sintilimab; Granulocyte-Macrophage Colony-Stimulating Factor; HMPL-013

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): hypofractionation radiotherapy combined with sintilimab,GM-CSF and Fruquintinib in the third-line or above treatment of MSS Metastatic Colorectal Carcinoma(mCRC)
  Interventions: Radiation: hypofractionation Radiotherapy; Drug: sintilimab; Drug: GM-CSF; Drug: Fruquintinib

INTERVENTIONS:
Radiation: hypofractionation Radiotherapy — Patients will receive radiation to the target lesion at a dose of 5Gy, 5 fractions a week, or a dose of 8Gy, 3 fractions a week. The course last once or twice depending on the investigator.
  Other Names: Radiotherapy
Drug: sintilimab — 200 mg per IV infusion every 21 days until disease progression or participant withdrawal from study or last for two years
  Other Names: IBI308
Drug: GM-CSF — 200µg given 7-14 days(until WBC≥40x109/L), every 21 days until disease progression or participant withdrawal from study or last for two years.
  Other Names: Human Granulocyte
Drug: Fruquintinib — Fruquintinib will be given 5mg qd for 2 weeks on and 1 week off, Q3W.
  Other Names: Elunate

SUMMARY:
To evaluate the clinical efficacy and safety of hypofractionation radiotherapy combined with sintilimab，GM-CSF and Fruquintinib in Patients With MSS Metastatic Colorectal Carcinoma (mCRC)

DETAILED DESCRIPTION:
Condition or disease:MSS Metastatic Colorectal Carcinoma (mCRC)

Phase:Phase 2

Intervention/treatment:

Radiation: hypofractionation radiotherapy

Drug: sintilimab, GM-CSF , Fruquintinib

ELIGIBILITY:
Inclusion Criteria:

* Assigned informed consent
* Age: 18-80 years
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-3
* Histological or cytological documentation of adenocarcinoma of the colon or rectum MSS metastatic colorectal cancer(CRC) checked by IHC or PCR.
* Patients must have failed at least two lines of prior treatment
* Patients must have not previously received anti-programmed death-1 (PD-1) or its ligand (PD-L1) antibody, anti-cytotoxic T lymphocyte-associated antigen 4 (cytotoxic T-lymphocyte-associated Protein 4, CTLA-4) antibody or other drug/antibody that acts on T cell costimulation or checkpoint pathways.
* Patients must have not previously received Fruquintinib.
* Life expectancy of at least 3 months
* At least 1 measurable disease according to Response Evaluation Criteria in Solid --Tumors (RECIST) criteria, version 1.1.is necessary.
* Controlled hypertension.
* Adequate bone marrow, liver and renal function as assessed by the laboratory required by protocol.
* Women of childbearing age must be negative in pregnancy test. Fertile female and male patients agree to use effective contraceptive methods during the study and within 6 months post to the last dose, such as double barrier contraception, condoms, oral or injection contraceptives, intrauterine devices, abstinence, etc. All female patients will be considered fertile unless the female patient has natural menopause or has undergone artificial menopause or sterilization (hysterectomy, bilateral appendage resection).

Exclusion Criteria:

* Patients with MSI-H / dMMR metastatic colorectal cancer(CRC);
* Uncontrollable malignant pleural effusion, ascites or pericardial effusion (defined as ineffectively controlled by diuresis or puncture drainage judged by investigators);
* Clinically significant abnormal electrolyte abnormality as judged by investigators;
* Clinically significant liver disease, including active viral hepatitis [HBsAg and/or HbcAb is positive and HBV (hepatitis B virus) DNA > 10000 copies/ mL or > 2000 IU/mL; HCV (hepatitis C virus) antibody positive and HCV RNA > 1000 copies/ mL], or other active hepatitis, clinically significant moderate to severe cirrhosis;
* Central nervous system (CNS) metastasis in previous or screening is excluded ,except CNS without clinical symptom or stable period ≥4 weeks after treatment ;
* Patients with evidence or history of propensity to hemorrhage within 3 months prior to first dosing, regardless of severity(such as melena, hematemesis, hemoptysis, bloody stools）；
* History of arterial thrombosis within 6 months; Patients with history of deep vein thrombosis (DVT) are eligible as long as they have received or are receiving appropriate anticoagulation therapy.
* Uncontrolled hypertension. (Systolic blood pressure 150 mmHg or diastolic pressure 90 mmHg despite optimal medical management).
* Radical radiotherapy within 4 weeks prior to first dosing;
* Patients have dysphagia;
* History of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, severe impairment of the lung function, etc., which may interfere with the detection and treatment of suspected drug-related lung toxicity, except radiation pneumonitis in the radiation treatment area;
* Confirmed human immunodeficiency virus (HIV) infection or confirmed syphilis; Patients have high risk of bleeding events such as unhealed wounds, ulcers, fractures,or. patients have active ulcer of stomach and duodenum, ulcerative colitis and other digestive tract diseases or unresectable tumors with active bleeding, or other conditions that may cause gastrointestinal bleeding and perforation, as judged by investigators;
* The adverse events due to previous anti-tumor therapy has not recovered to ≤ CTCAE Grade 1, except alopecia and peripheral neurotoxicity with ≤ CTCAE grade 2 caused by platinum chemotherapy;
* Patients with active infection and still need systemic treatment;
* Steroids (more than 10 mg/day prednisone or other equivalent hormones) or other immunosuppressive agents for systemic therapy within 4 weeks prior to first dosing, except nasal spray, inhaled or other topical use of steroid (i.e. no more than 10mg/day prednisone or equivalent doses of other corticosteroids);
* Any live or attenuated live vaccine within 4 weeks prior to first dosing;
* Major surgeries within 4 weeks prior to first dosing;
* Any anti-tumor traditional Chinese medicine taken within 2 weeks prior to first dosing;
* History of allergies to any ingredient of Sintilimab or Fruquintinib or GM-CSF;
* Participating in other interventional clinical studies within 4 weeks;
* Female patients with pregnancy or breastfeeding;
* Urine routines show urine protein≥ ++, or urine protein quantity≥ 1.0 g during 24 hours；
* History of any active autoimmune disease or autoimmune disease, including but not limited to interstitial pneumonia, uveitis, inflammatory bowel disease, hepatitis, pituitary inflammation, vasculitis, systemic lupus erythematosus, etc. (except patients with hypothyroidism that can be controlled only by hormone replacement therapy and patients with type I diabetes who only need insulin replacement therapy);
* Patients with uncontrolled epilepsy, central nervous system disease, or mental disorders whose clinical severity, as determined by the investigator, may prevent the signing of the informed consent or any condition by which investigators judge patients not suitable to participate in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2022-03-25 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 2 years
  Defined as the time from the date of the first dose of treatment to the date of the first documentation of disease progression or death, whichever occurs first.
  Progression-free survival (PFS) according to Response Evaluation Criteria in Solid Tumours (RECIST) version. 1.1, and immune-related (ir) RECIST

SECONDARY OUTCOMES:
Objective response rate | 1 year
  Objective response rate (ORR) according to Response Evaluation Criteria in Solid Tumours (RECIST) version. 1.1, and immune-related (ir) RECIST
Disease Control Rate（DCR） | 1 year
  Disease Control Rate（DCR）according to Response Evaluation Criteria in Solid Tumours (RECIST) version. 1.1, and immune-related (ir) RECIST
Duration of Response(DOR) | 1 year
  Duration of Response(DOR) according to Response Evaluation Criteria in Solid Tumours (RECIST) version. 1.1, and immune-related (ir) RECIST
Overall survival (OS) | 2 years
  Defined as the time from the date of the first dose of treatment until the date of death due to any cause.
Safety:Percentage of Participants With Adverse Events (AEs) | Up to 30 days after the last cycle of per-protocol treatment and 90 days after last dose of treatment
  Percentage of Participants With Adverse Events (AEs) Number of participants with adverse events occurring up to 30 days after the last administration are evaluated and graded according to the National Cancer Institute Common Terminology Criteria (NCI CTCAE) for Adverse Events, version 5.01

CONTACTS AND LOCATIONS:
Overall Officials: Mingquan Cai, Principal Investigator — The First Affiliated Hospital of Xiamen University; Xiyi Liao, Principal Investigator — The First Affiliated Hospital of Xiamen University
Locations (1):
- The First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No